CLINICAL TRIAL: NCT04854720
Title: Clinical Efficacy of Different Fissure Sealant Materials in the Newly Erupted Non-Carious First Permanent Molars: A Randomized Controlled Clinical Trial
Brief Title: Clinical Efficacy of Different Fissure Sealant Materials in the Newly Erupted Non-Carious First Permanent Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Merve AKCAY, Assoc. Prof. Dr., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-TDU-DİŞF-0050
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Fissure Sealant
Keywords: Conventional glass ionomer; fissure sealant; giomer; laser fluorescence; newly erupted teeth; resin modified glass ionomer

STUDY DESIGN:
Intervention Model Description: randomized controlled, three-arm parallel, single-blinded, split-mouth clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization was performed by a computer-generated random sorting sequence (sealed in opaque envelopes that sequentially numbered randomly selected through).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Fuji II LC-Fuji Triage) (Experimental): In Group 1, newly erupted mandibular permanent first molars were sealed with resin-modified glass ionomers containing fissure sealant material (Fuji® II LC, GC Corporation, Tokyo, Japan) (test 1). The other first molars were sealed with glass ionomers containing fissure sealant material (Fuji Triage®, GC Corporation, Tokyo, Japan) (control).
  Interventions: Device: Fuji® II LC CAPSULE; Device: Fuji Triage® CAPSULE
- Group 2 (Clinpro XT Varnish-Fuji Triage) (Experimental): In Group 2, newly erupted mandibular permanent first molars were sealed with resin-modified glass ionomers containing fissure sealant material (Clinpro™ XT Varnish, 3M ESPE, St. Pauls, Miniapolis, MN, USA) (test 2). The other first molars were sealed with glass ionomers containing fissure sealant material (Fuji Triage®, GC Corporation, Tokyo, Japan) (control).
  Interventions: Device: Clinpro™ XT Varnish; Device: Fuji Triage® CAPSULE
- Group 3 (Beautiful Flow- Fuji Triage) (Experimental): In Group 3, newly erupted mandibular permanent first molars were sealed with Giomer containing fissure sealant material (Beautifil Flow, Shofu, Kyoto, Japan) (test 3). The other first molars were sealed with glass ionomers containing fissure sealant material (Fuji Triage®, GC Corporation, Tokyo, Japan) (control).
  Interventions: Device: Beautifil Flow; Device: Fuji Triage® CAPSULE

INTERVENTIONS:
Device: Fuji® II LC CAPSULE — Fuji® II LC is a resin modified glass ionomer contained, fluoride releasing and light-cured material. Since the product is tolerant to moisture and saliva, it's used for fissure sealant of newly erupted teeth.
  Test 1 newly erupted first permanent molars were cleaned with a pumice paste using a bristle brush and isolated with cotton rolls. Then, 20% cavity conditioner was applied to all surfaces of the tooth for 10 seconds.The tooth surface was rinsed with water and dried. Thereafter, Fuji® II LC was applied to the pits and fissures on the tooth surface using a brush. Then, the varnish was applied and cured according to the manufacturer's instructions.
  Other Names: Fuji® II LC CAPSULE, GC Corporation, Tokyo, Japan
  Arms: Group 1 (Fuji II LC-Fuji Triage)
Device: Clinpro™ XT Varnish — Clinpro™ XT Varnish is a resin modified glass ionomer containing, fluoride-releasing, light-cured varnish. Since the product is tolerant to moisture and saliva, it is used for fissure sealant of newly erupted teeth. The product can be recharged with fluoride using fluoride-containing products.
  Test 2 newly erupted first permanent molars were cleaned with a pumice paste using a bristle brush and isolated with cotton rolls. Then, 35% phosphoric acid was applied to all surfaces of the tooth for 15 seconds.Then the tooth surface was rinsed with water and dried. Thereafter, Clinpro™ XT Varnish was applied in compliance with the manufacturers' instructions.
  Other Names: Clinpro™ XT Varnish, 3M ESPE, St. Pauls, Miniapolis, MN, USA
  Arms: Group 2 (Clinpro XT Varnish-Fuji Triage)
Device: Beautifil Flow — Beautiful Flow is a Giomer contained, fluoride releasing and light cured material. The product contains pre-reacted glass ionomer particles (PRG). It is a high water resistant material. It is used for fissure sealant.
  Test 3 newly erupted first permanent molars were cleaned with a pumice paste using a bristle brush and isolated with cotton rolls. Then, 7% phosphoric acid was applied to all surfaces of the tooth for 10 seconds. Then the tooth surface was rinsed with water and dried. Afterwards, a two-stage self-etch adhesive system was applied. Thereafter, Beautiful Flow was applied in compliance with the manufacturers' instructions.
  Other Names: Beautifil Flow, Shofu, Kyoto, Japan
  Arms: Group 3 (Beautiful Flow- Fuji Triage)
Device: Fuji Triage® CAPSULE — Fuji Triage® is a new generation glass ionomer containing with low viscosity, high fluoride content and light curing materials. Since the product is tolerant of moisture and saliva, it is used for fissure sealant of newly erupted teeth.
  Control newly erupted first permanent molars were cleaned with a pumice paste using a bristle brush and isolated with cotton rolls. Then, 20% cavity conditioner was applied to all surfaces of the tooth for 10 seconds.Then the tooth surface was rinsed with water and dried. Thereafter,Fuji Triage® was applied to the pits and fissures on the tooth surface using a brush. Thereafter, the varnish was applied and cured according to the manufacturer's instructions.
  Other Names: Fuji Triage® CAPSULE, GC Corporation, Tokyo, Japan

SUMMARY:
The aim of this study is to compare the clinical retention rates, marginal adaptation, marginal discoloration and secondary caries formation of two different types of resin-modified glass ionomers (Fuji® II LC; Clinpro™ XT Varnish) and giomer-containing fissure sealant materials (Beautifil Flow) with glass ionomer-containing fissure sealant material (Fuji Triage®) used on newly erupted non-carious first permanent molars as a fissure sealant.

The study included 384 teeth belonging to 182 children, aged between 5 to 9 years old, who have two newly erupted mandibular permanent first molars.

DETAILED DESCRIPTION:
Firstly, patients were randomly allocated to three main groups: Group 1; Fuji II LC/Fuji Triage (Control) (62 patients), Group 2; Clinpro XT Varnish/Fuji Triage (Control) (60 patients), Group 3; Beautifil Flow/Fuji Triage (Control) (60 patients). After clinical applications, all samples were evaluated in terms of retention, marginal adaptation, marginal discoloration and secondary caries formation using modified USPHS criteria in 6th, 12th and 18th months. Also samples were evaluated in terms of remineralization effect using the laser fluorescence method. Evaluations on occlusal and buccal surfaces were performed separately.

ELIGIBILITY:
Inclusion Criteria:

* Children who have two newly erupted non-carious mandibular permanent first molars that fissure sealant is indicated,
* Newly erupted first permanent molars show scores of 0 (Sound tooth surface)-1(First visual change in enamel) according to ICDAS II,
* Newly erupted first permanent molars show scores between 0-13 by using DIAGNOdent device,
* Children who haven't any systemic disease that prevents the application,
* Cooperative children who allowed the clinical applications.

Exclusion Criteria:

* Teeth with proximal and initial caries,
* Teeth with applied fissure sealant,
* Teeth with developmental defects such as hypoplasia and restorations,
* Non-cooperative children who don't allow the clinical applications,
* Children and parents who denied the participation in the follow-up appointments.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
The assessment of clinical retention rates of fissure sealants applied to newly erupted permanent first molars. | 18 months after the clinical applications
  The primary outcome of the study was the assessment of clinical retention rates at 18th months.
The assessment of marginal adaptation rates of fissure sealants applied to newly erupted permanent first molars. | 18 months after the clinical applications
  The primary outcome of the study was the assessment of marginal adaptation rates at 18th months.
The assessment of marginal discoloration rates of fissure sealants applied to newly erupted permanent first molars. | 18 months after the clinical applications
  The primary outcome of the study was the assessment of marginal discoloration rates at 18th months.
The assessment of secondary caries rates of fissure sealants applied to newly erupted permanent first molars. | 18 months after the clinical applications
  The primary outcome of the study was the assessment of secondary caries rates at 18th months.

SECONDARY OUTCOMES:
The assessment of remineralization capacity using DIAGNOdent device | 18 months after the clinical applications
  The secondary outcome of the study was the assessment of remineralization capacity using DIAGNOdent, at 18th months.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Akcay, assoc. prof., Study Chair — Izmir Katip Celebi Uni
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No